CLINICAL TRIAL: NCT00688467
Title: A Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy and Safety of SCH 527123 in Subjects With Allergen-Induced Asthma
Brief Title: Efficacy and Safety of Navarixin (SCH 527123) in Participants With Allergen-Induced Asthma (P05363)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P05363; MK-7123-016 (Other: Merck protocol number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Asthma
Keywords: Neutrophilic Asthma
MeSH Terms: conditions — Asthma | interventions — navarixin; 2-hydroxy-N,N-dimethyl-3-(2-((1-(5-methylfuran-2-yl)propyl)amino)-3,4-dioxocyclobut-1-enylamino)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navarixin → Placebo (Experimental): Navarixin 30 mg capsule to be taken once daily in the morning for 10 days in Treatment Period 1, followed by a 2-4 week washout period, followed by matching placebo capsule to be taken once daily in the morning for 10 days in Treatment Period 2
  Interventions: Drug: Navarixin; Drug: Placebo
- Placebo → Navarixin (Experimental): Matching placebo capsule to be taken once daily in the morning for 10 days in Treatment Period 1, followed by a 2-4 week washout period, followed by navarixin 30 mg capsule to be taken once daily in the morning for 10 days in Treatment Period 2
  Interventions: Drug: Navarixin; Drug: Placebo

INTERVENTIONS:
Drug: Navarixin — 30 mg capsule to be taken once daily in the morning for 10 days during Treatment Period 1 or Treatment Period 2
  Other Names: SCH 527123
Drug: Placebo — Matching capsule to be taken once daily in the morning for 10 days during Treatment Period 1 or Treatment Period 2

SUMMARY:
Evaluation of treatment in participants with mild asthma.

DETAILED DESCRIPTION:
To evaluate the effect of navarixin (MK-527123, SCH 527123) treatment on allergen-induced late asthmatic response (LAR) in participants with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 to 65 years of age of any race.
* Has mild, stable, allergic asthma as defined by American Thoracic Society criteria.
* Has history of episodic wheezing and shortness of breath.
* Has Forced Expiratory Volume in 1 second (FEV1) of at least 70% of predicted at Screening and within 10% of preallergen screening value at both baselines.
* Has positive methacholine challenge at Screening. Methacholine challenges are considered positive if decreases of at least 20% in the FEV1 occur at a concentration of less than or equal to 16 mg/mL.
* Baseline methacholine PC20 (concentration that initiated a 20% fall in FEV1) must be within 1 doubling concentration of the preallergen screening PC20 to enter treatment.
* Has positive skin-prick test to common allergens (cat, dust mite, grass, pollen).
* Has a positive Early Asthmatic Response of >=20% fall in FEV1 measured from the FEV1 immediately prior to challenge, and Late Asthmatic Response of >=15% fall in FEV1 from the FEV1 measured immediately prior to challenge during Screening period.
* Has been free from asthma exacerbation for at least 4 weeks before Screening. An exacerbation is defined as an occurrence of any clinical deterioration of asthma that requires emergency treatment, hospitalization due to asthma, or treatment with additional medication, as judged by the clinical investigator.
* Has been free from relevant seasonal allergen exposure for at least 4 weeks before the study and be able to remain so for the duration of the study.
* Has a current nonsmoking status. If previous smokers, cumulative smoking history must be fewer than 10 pack-years (pack-year=20 cigarettes smoked daily for 1 year). Previous smokers must not have smoked within 1 year before Screening.
* Is willing to give written informed consent to participate in the study.
* Has the ability to comply with the dosing regimen, to adhere to the visit schedule, and to participate in all treatment procedures, including sputum induction.
* Female participant of childbearing potential must have a negative serum pregnancy tests (human chorionic gonadotropin; hCG) at Screening and must use a medically acceptable, highly effective, adequate form of birth control (ie, failure rate <1% per year when used consistently and correctly) prior to Screening and agrees to continue using it while in the study (Screening and Treatment Periods). Medically acceptable, highly effective forms of birth control include hormonal implants, oral contraceptives, hormonal patches, intravaginal ring, medically acceptable prescribed intrauterine devices (IUDs), and a monogamous relationship with a male partner who has had a vasectomy. A female participant who is not of childbearing potential must have a medical record of being surgically sterile (eg, hysterectomy, tubal ligation), or be at least 1 year postmenopausal. Absence of menses for at least 1 year will indicate that a female is postmenopausal. A female participant should be encouraged to continue using a highly effective method of birth control for 30 days following the end of treatment.
* Participants, if male and sexually active with women of childbearing potential, must agree to use an adequate form of contraception for the duration of the study and to have sexual relations with only those women who use a highly effective birth control method.
* Clinical laboratory tests (complete blood count [CBC], blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator/sponsor.

Exclusion Criteria:

* Has had a diagnosis of chronic obstructive pulmonary disease (COPD) or any other clinically relevant lung disease (eg, cystic fibrosis, pulmonary fibrosis, bronchiectasis) other than mild allergic asthma, or has a history of having been intubated.
* Has had a worsening of a respiratory tract infection within 4 weeks before Screening.
* Has had any clinically significant abnormality; history of clinically significant hypotensive episodes of fainting, dizziness, or lightheadedness; history or symptoms of cardiovascular disease; significant neurologic disease; or hematologic abnormality, including coagulopathy; or has a medication regimen or clinically relevant medical condition other than asthma that may interfere with the effect of study medication.
* Had a peripheral blood neutrophil (PBN) count of <3 × 10^9/L at the Screening Visit.
* Has an allergy/sensitivity to the study drug or its excipients.
* Is pregnant, breast-feeding, or intends to become pregnant during the study.
* Has used any investigational drug within 30 days or 5 half-lives of Screening.
* Is presently participating in any other clinical study.
* Is part of the staff personnel directly involved with this study
* Is a family member of the investigational study staff.
* Has received any treatment prohibited by the protocol (Table 3), or any medication that may interfere with the effect of the study medication more recently than the indicated washout period prior to Screening, or must continue to receive the prohibited treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05363&kw=P05363&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Navarixin → Placebo | Placebo → Navarixin
Started | 9 | 10
Completed | 7 | 8
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Did not meet protocol eligibility | 0 | 1
Period: Treatment Period 2
Arm/Group | Navarixin → Placebo | Placebo → Navarixin
Started | 7 | 8
Completed | 7 | 6
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Navarixin → Placebo | Placebo → Navarixin | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (12.0) | 24.9 (4.0) | 29.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve From 3 to 7 Hours (AUC3-7hr) After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: This is a measure of the Late Asthmatic Response (LAR) between 3 and 7 hours after allergen challenge. Allergen challenge was administered 1 hour after the ninth daily dose of study drug in each treatment period. Baseline FEV1 was defined as the prechallenge FEV1 in the treatment period. A percent change >0 indicates a fall in FEV1 after allergen challenge. The reported standard deviations (SDs) are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups. The pooled SD values were used in the calculation of test statistics to assess treatment differences (p-value generation).
Time Frame: Baseline and between 3 and 7 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods
Measure: Least Squares Mean (Standard Deviation); unit: Percent change from baseline
Groups:
- Navarixin: Navarixin 30 mg capsule to be taken by mouth once daily in the morning for 10 days
- Placebo: Placebo 30 mg capsule to be taken by mouth once daily in the morning for 10 days
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 13 | 13
Percent change from baseline | 26.225 (27.377) [-16.977 to 94.929] | 35.427 (27.377) [-17.726 to 92.784]
Statistical Analysis 1: Comparison: Navarixin vs Placebo; Test type: Superiority or Other; p = 0.411, ANOVA; 100 * (placebo - navarixin) / placebo = 26.0, Standard Deviation 27.377

2. Secondary Outcome: Maximum Change From Baseline in FEV1 During the LAR Following 9 Days of Pretreatment With Navarixin
Description: Allergen challenge was administered 1 hour after the ninth daily dose of study drug in each treatment period. Baseline FEV1 was defined as the prechallenge FEV1 in the treatment period. The LAR was 3 to 7 hours after allergen challenge. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups. The pooled SD values were used in the calculation of test statistics to assess treatment differences (p-value generation).
Time Frame: Baseline and between 3 and 7 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 13 | 13
Liters | 0.438 (0.306) | 0.571 (0.306)
Statistical Analysis 1: Comparison: Navarixin vs Placebo; Test type: Superiority or Other; p = 0.292, ANOVA; 100 * (placebo - navarixin) / placebo = 23.3, Standard Deviation 0.306

3. Secondary Outcome: Change in Concentration of Methacholine That Initiated a 20% Reduction in FEV1 From 24 Hours Before (Baseline) to 24 Hours After Allergen Challenge
Description: This is a measure of allergen-induced changes in airway responsiveness to methacholine. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and 24 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods
Measure: Least Squares Mean (Standard Deviation); unit: Log methacholine (mg/mL)
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 13 | 13
Log methacholine (mg/mL) | -0.154 (0.205) | -0.161 (0.205)

4. Secondary Outcome: Percent Change From Baseline in FEV1 Area Under the Curve From 0 to 2 Hours (AUC0-2hr) After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: This is a measure of Early Asthmatic Response (EAR) between 0 to 2 hours after allergen challenge. Allergen challenge was administered 1 hour after the ninth daily dose of study drug in each treatment period. A percent change >0 indicates a reduction in FEV1 from before to after allergen challenge. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups. The pooled SD values were used in the calculation of test statistics to assess treatment differences (p-value generation).
Time Frame: Baseline and between 0 to 2 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods
Measure: Least Squares Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 13 | 13
Percent change from baseline | 35.924 (16.261) | 35.325 (16.261)
Statistical Analysis 1: Comparison: Navarixin vs Placebo; Test type: Superiority or Other; p = 0.927, ANOVA; 100 * (placebo - navarixin) / placebo = -1.7, Standard Deviation 16.261

5. Secondary Outcome: Maximum Percent Change From Baseline in FEV1 During the Early Asthmatic Response Following 9 Days of Pretreatment With Navarixin
Description: Allergen challenge was administered 1 hour after the ninth daily dose of study drug in each treatment period. The EAR was 0 to 2 hours after allergen challenge. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups. The pooled SD values were used in the calculation of test statistics to assess treatment differences (p-value generation).
Time Frame: Baseline and between 0 to 2 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods
Measure: Least Squares Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 13 | 13
Percent change from baseline | 30.872 (7.398) | 32.251 (7.398)
Statistical Analysis 1: Comparison: Navarixin vs Placebo; Test type: Superiority or Other; p = 0.645, ANOVA; 100 * (placebo - navarixin) / placebo = 4.3, Standard Deviation 7.398

6. Secondary Outcome: Change From Baseline in Sputum Neutrophils After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: Induced sputum samples were collected via the nebulized method. Baseline values were determined at 24 hours before allergen challenge in each treatment period. Sputum neutrophils were measured as percent of total white blood cells. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and 7 and 24 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods and were able to produce evaluable sputum samples
Measure: Least Squares Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 4 | 5
Percent change from baseline
  7 hours after allergen challenge (n=3, n=4) | -45.043 (31.188) | -8.189 (31.188)
  24 hours after allergen challenge (n=4, n=5) | -40.412 (10.302) | 7.057 (10.302)

7. Secondary Outcome: Change From Baseline in Peripheral Blood Eosinophil Count After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: Baseline values were determined at 24 hours before allergen challenge in each treatment period. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and 7 and 24 hours after allergen challenge
Population: The population analyzed included all participants who completed both treatment periods and had evaluable blood samples available
Measure: Least Squares Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 13 | 13
Percent change from baseline
  7 hours after allergen challenge (n=11, n=12) | -0.066 (0.106) | -0.029 (0.106)
  24 hours after allergen challenge (n=13, n=13) | 0.034 (0.089) | 0.078 (0.089)

8. Secondary Outcome: Change From Baseline in Sputum Interleukin 8 (IL-8) After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: Induced sputum samples were to be collected via the nebulized method. IL-8 level was measured in the sputum supernatant. Baseline values were determined at 24 hours before allergen challenge in each treatment period. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and 7 and 24 hours after allergen challenge
Population: as for outcome 6
Measure: Least Squares Mean (Standard Deviation); unit: pg/mL
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 6 | 6
pg/mL
  7 hours after allergen challenge (n=6, n=4) | -1746.5 (7167.68) | 18136.2 (7167.68)
  24 hours after allergen challenge (n=6, n=6) | -856.66 (8149.08) | 13195.2 (8149.08)

9. Secondary Outcome: Change From Baseline in Sputum Neutrophil Elastase After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: Induced sputum samples were to be collected via the nebulized method. Neutrophil elastase activity was measured in the sputum supernatant as milli units/mL (mU/mL). Baseline values were determined at 24 hours before allergen challenge in each treatment period. The reported SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and 7 and 24 hours after allergen challenge
Population: as for outcome 6
Measure: Least Squares Mean (Standard Deviation); unit: mU/mL
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 6 | 6
mU/mL
  7 hours after allergen challenge (n=6, n=4) | -254.92 (380.316) | 230.416 (380.316)
  24 hours after allergen challenge (n=6, n=6) | -166.27 (303.402) | 2.264 (303.402)

10. Secondary Outcome: Change From Baseline in Sputum Myeloperoxidase (MPO) Level After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: Induced sputum samples were to be collected via the nebulized method. MPO level was measured in the sputum supernatant.
Time Frame: Baseline and 7 and 24 hours after allergen challenge
Population: MPO level was not analyzed because too few evaluable samples were collected
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Sputum Eosinophil Cationic Protein (ECP) Level After Allergen Challenge Following 9 Days Pretreatment With Navarixin
Description: Induced sputum samples were to be collected via the nebulized method. ECP level was measured in the sputum supernatant.
Time Frame: Baseline and 7 and 24 hours after allergen challenge
Population: ECP level was not analyzed because too few evaluable samples were collected
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to study drug. AEs were reported based on the study drug taken at the time of the event.
Time Frame: Up to 48 days
Population: The population analyzed included all participants who received study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 16 | 17
Participants | 8 | 8

13. Secondary Outcome: Number of Participants Discontinued From the Study Because of an Adverse Event
Description: An AE is any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to study drug. Discontinuations due to an AE are reported based on the study drug taken at the time of the event.
Time Frame: Up to 48 days
Population: The population analyzed included all participants who received study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 16 | 17
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 48 days (the day of the last dose of study drug in Treatment Period 2)
Description: Adverse events were collected for all participants who received >=1 dose of study drug in either treatment period. Adverse events were reported based on the study drug taken at the time of the event.
Arm/Group | Navarixin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/17
Other Adverse Events (participants affected / at risk) | 8/16 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin (N=16) | Placebo (N=17)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin (N=16) | Placebo (N=17)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.